CLINICAL TRIAL: NCT05951569
Title: An Observational Study of Adults With Type 2 Diabetes Using the Community-Derived Open-Source Automated Insulin Delivery Loop System
Brief Title: Loop T2D Observational Study
Status: Completed | Type: Observational
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Embecta Medical (Unknown); Tidepool Project (Unknown)
Responsible Party: Sponsor
Other Study IDs: T2D Loop
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Loop; Type 2 Diabetes; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Autoimmune Diseases; Immune System Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Autoimmune Diseases; Immune System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Community-Derived Open-Source Automated Insulin Delivery Loop System — The Loop System consists of an insulin pump and a Dexcom CGM. The system includes an iPhone with the Loop app and a RileyLink to communicate between the pump and iPhone. An Apple Watch may optionally be used with the system.

SUMMARY:
An observational study to collect data on the efficacy, safety, usability, and quality of life/psychosocial effects of the community-derived OS-AID Loop System on adults with type 2 diabetes.

DETAILED DESCRIPTION:
The study will include adults with type 2 diabetes in the United States, with a recruitment goal of a maximum of 100 participants. Data to be collected to address the study objective will include CGM metrics; HbA1c; insulin delivery data; carbohydrate data; activity data from HealthKit; self-reported adverse events (e.g., severe hypoglycemia, diabetic ketoacidosis, hospitalizations); self-reported device issues; and user experience/treatment satisfaction surveys.

Follow-up data will be collected on a monthly basis as long as the study is continuing and participants are still using Loop.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Age ≥18 years old
* Currently using any version of Loop other than v3.0.0 or planning to start using any version of Loop other than v3.0.0 Loop within the next 30 days
* Willing and able to provide informed consent and to complete surveys and provide the device data that are part of the protocol
* Resident of the US
* English speaking/reading
* Access to email/phone

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with type 2 diabetes using the community-derived open-source automated insulin delivery Loop system.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
Measure of Loop Safety by Self-Report of Diabetic Ketoacidosis (DKA) Events | Up to 3 months
  Number of DKA events and event outcomes. DKA events are defined as hospitalization with documentation of arterial blood pH <7.30 or venous pH <7.24 or serum bicarbonate (or CO2) <15.
Measure of Loop Safety by Self-Report of Severe Hypoglycemic Events | Up to 3 months
  Number of severe hypoglycemic events and event outcomes. Severe hypoglycemia is defined as low blood sugar that affected the individual's ability to think such that they were unable to treat themselves and needed assistance from someone else. The individual may or may not have lost consciousness.
Measure of Loop Safety by Self-Report of Hospitalization Events | Up to 3 months
  Number of hospitalizations

OTHER OUTCOMES:
Loop T2D Baseline General Data Collection | Enrollment
  Self-report participant's basic information. No scale provided, variable responses.
Loop T2D Follow-up Survey | Monthly up to 3 months
  Self-report of participant's use of Loop and Loop related features. No scale provided, variable responses.
HbA1c | Enrollment, Monthly up to 3 months
  Self-report

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Bauza, PhD, MPH, Principal Investigator — Jaeb Center for Health Research
Locations (1):
- Jaeb Center for Health Research, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lum JW, Bailey RJ, Barnes-Lomen V, Naranjo D, Hood KK, Lal RA, Arbiter B, Brown AS, DeSalvo DJ, Pettus J, Calhoun P, Beck RW. A Real-World Prospective Study of the Safety and Effectiveness of the Loop Open Source Automated Insulin Delivery System. Diabetes Technol Ther. 2021 May;23(5):367-375. doi: 10.1089/dia.2020.0535. Epub 2021 Apr 12. PMID 33226840
- [Derived] Bauza C, Kanapka LG, Greene E, Lal RA, Arbiter B, Beck RW. Use of the Community-Derived Open-Source Automated Insulin Delivery Loop System in Type 2 Diabetes. Diabetes Technol Ther. 2024 Jul;26(7):494-497. doi: 10.1089/dia.2023.0569. Epub 2024 Apr 8. PMID 38386434